CLINICAL TRIAL: NCT05992467
Title: WECARE: A mHealth Intervention to Enhance Caregiving Mastery Among Chinese American Dementia Caregivers
Brief Title: WECARE: A Behavioral Intervention for Dementia Caregivers
Acronym: WECARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Mason University (Other)
Responsible Party: Principal Investigator, Y. Alicia Hong, Professor, George Mason University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: George Mason University
Record Dates: First submitted 2023-07-06; First posted 2023-08-15 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Caregiver Burden; Caregiver Stress Syndrome
MeSH Terms: conditions — Caregiver Burden | interventions — Caregivers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- WECARE (Experimental): Participants will first complete a baseline survey online, then subscribe to the WECARE official account on their own WeChat accounts and begin receiving the 7-week interactive and personalized program. The program content includes short video clips, pictorial messages, and audio recordings. Each week, the WECARE program is focused on a theme aimed to increase participants' caregiving mastery, enhance self-care, and improve psychosocial wellbeing. Four weeks after the intervention or 11 weeks after the baseline, participants will complete a follow-up survey online.
  Interventions: Behavioral: Wellness Enhancement for Caregivers (WECARE)

INTERVENTIONS:
Behavioral: Wellness Enhancement for Caregivers (WECARE) — WECARE behavioral intervention is guided by behavioral theories aimed to increase participants' caregiving mastery, enhance self-care, and improve psychosocial wellbeing. Participants will receive multimedia content on their WeChat account on cellphone or tablet, including short video clips, pictorial messages, short articles, and audio recordings 6 days a week, for 7 weeks.

SUMMARY:
This study aims to pilot test a culturally tailored behavioral intervention called "WECARE" to enhance caregiving mastery and improve psychosocial wellbeing of Chinese American family caregivers of persons with Alzheimer's Disease and related dementia.

DETAILED DESCRIPTION:
The investigators propose to test a culturally tailored mHealth behavioral intervention to enhance caregiving mastery and improve psychosocial wellbeing among Chinese American family caregivers of persons living with Alzheimer's Disease and related dementia. This intervention, Wellness Enhancement for Caregivers (WECARE), will be delivered via WeChat, a social media app highly popular among Chinese Americans. About 45 participants will be recruited for the pilot test. Participants will complete a baseline survey, receive 7-week WECARE program on their WeChat accounts, complete a follow-up survey 12 weeks after the baseline, and then a qualitative interview on Zoom.

ELIGIBILITY:
Inclusion Criteria:

1. 21 years or older,
2. self-identified as Chinese or Chinese American,
3. speak and read Chinese (Mandarin or Cantonese),
4. own a smartphone and use WeChat,
5. living in Washington DC metropolitan, and
6. currently care for a family member with ADRD and provide care for at least 10 hours a week.

Exclusion Criteria:

1. do not read or speak Chinese,
2. care-recipient is in hospice care or have a life expectancy less than 6 months,
3. signs of severe intellectual deficits or psychotic disorders, or
4. unable to provide informed consent.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Efficacy of behavioral intervention in change from baseline in depressive symptoms | Baseline (before the intervention) and follow-up (week 11-12, or 4-5 weeks after the intervention
  The baseline and follow-up differences in depressive symptoms will be assessed. Depressive symptoms will be measured by the CES-D, a 20-item survey instrument. The total score will be calculated to quantify depressive symptoms. The baseline and follow-up differences in the scores will be calculated.

SECONDARY OUTCOMES:
Efficacy of behavioral intervention in change from baseline in caregiving burden | Baseline (before the intervention) and follow-up (week 11-12, or 4-5 weeks after the intervention
  The baseline and follow-up differences in caregiving burden will be assessed. Caregiving burden will be measured by the Zarit Burden Interview, a 12-item survey instrument. The total score will be calculated to quantify caregiving burden. The baseline and follow-up differences in the scores will be calculated.
Efficacy of behavioral intervention in change from baseline in life satisfaction | Baseline (before the intervention) and follow-up (week 11-12, or 4-5 weeks after the intervention
  The baseline and follow-up differences in life satisfaction will be assessed. Life satisfaction will be measured by the Life Satisfaction Scale, a 5-item survey instrument. The total score will be calculated to quantify life satisfaction. The baseline and follow-up differences in the scores will be calculated.

OTHER OUTCOMES:
Efficacy of behavioral intervention in change from baseline in caregiving mastery | Baseline (before the intervention) and follow-up (week 11-12, or 4-5 weeks after the intervention
  The baseline and follow-up differences in caregiving mastery will be assessed. Caregiving mastery will be measured by the Caregiving Mastery Scale, a 7-item survey instrument. The total score will be calculated to quantify caregiving mastery. The baseline and follow-up differences in the scores will be calculated.
Efficacy of behavioral intervention in change in care-recipient's problem behaviors | Baseline (before the intervention) and follow-up (week 11-12, or 4-5 weeks after the intervention
  The baseline and follow-up differences in care-recipient's problem behaviors will be assessed. Care-recipient's problem behaviors will be measured by a list of 20-item problem behaviors. The total score will be calculated to quantify the number of problem behaviors. The baseline and follow-up differences in the scores will be calculated.
Efficacy of behavioral intervention in change from baseline in positive aspect of caregiving | Baseline (before the intervention) and follow-up (week 11-12, or 4-5 weeks after the intervention.
  The baseline and follow-up differences in caregivers' positive aspects of caregiving will be measured by Positive Aspects of Caregiving Scale, a 9-item scale 5-point Likert scale from 0 to 4, with total scores ranging from 0 to 36, with higher score indicating more positive perception of caregiving. The baseline and follow-up differences in the scores will be calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- George Mason University, Fairfax, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
Given the small sample size, we will not make individual participant data available to the public.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After the investigators completes primary data collection and the first report from this trial is accepted for publication.
Access Criteria: Researchers will submit a request including the purpose of accessing the data and a data user agreement